CLINICAL TRIAL: NCT04469894
Title: Understanding Health Insurance Literacy and Challenges in Accessing Health Services in Niemann-Pick Disease Through the Eyes of Patients and Families
Brief Title: Health Insurance Literacy and Challenges in Accessing Health Services in Niemann-Pick
Status: Completed | Type: Observational
Sponsor: National Niemann-Pick Disease Foundation (Other)
Collaborators: Engage Health Inc. (Industry); Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Sponsor
Other Study IDs: NNPDF-BUR001
Record Dates: First submitted 2020-07-10; First posted 2020-07-14 (Actual); Last update posted 2020-10-06 (Actual); Status verified 2020-10

CONDITIONS: Niemann-Pick Diseases
MeSH Terms: conditions — Niemann-Pick Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (7):
- Niemann-Pick Type A: Also referred to as Infantile Neurovisceral ASMD
- Niemann-Pick Type A/B: Also referred to as Intermediate form or Chronic Neurovisceral ASMD
- Niemann-Pick Type B: Also referred to as Chronic Visceral ASMD
- Niemann-Pick Type C (Early Infantile): Onset at less than 2 years of age
- Niemann-Pick Type C (Late Infantile): Neurodegenerative form (late-infantile) onset at 2-6 years of age
- Niemann-Pick Type C (Juvenile): Neurodegenerative form (juvenile) onset at 6-15 years of age
- Niemann-Pick Type C (Adult): Psychiatric neurodegenerative form (adult) onset at greater than 15 years of age

SUMMARY:
This study is a US based qualitative PRO research study to document the health insurance literacy as well as the patient experience in Niemann-Pick as it relates to accessing desired care, services and medications for patients.

The outcome of this research will be used to inform various other workstreams as NNPDF works to assist families.

The core research objectives are to understand the following from Niemann-Pick patients and their families in the US

DETAILED DESCRIPTION:
This study is a US based qualitative PRO research study to document the health insurance literacy as well as the patient experience in Niemann-Pick as it relates to accessing desired care, services and medications for patients.

The outcome of this research will be used to inform various other workstreams as NNPDF works to assist families.

The core research objectives are to understand the following from Niemann-Pick patients and their families in the US;

* Level of health insurance literacy through assessment of health insurance terminology, and self-reported insights regarding information seeking, document literacy and cognitive skills
* If they have healthcare insurance, and if not, why not
* Types (including name) of insurance by which Niemann-Pick families are covered
* Information regarding Medicaid Waivers
* Attributes of insurance plans including, but not limited to;

  * Deductible amounts for individual and family
  * Out of pocket maximums for individual and family
  * Insurance premiums
  * Associated Health Savings Accounts
  * Associated Cost Sharing requirements
  * Services, drugs and assistive devices covered
* What the perceived out-of-pocket costs are for Niemann-Pick families (annually)
* When out-of-pocket maximums are perceived to be met for Niemann-Pick families
* Patient and HCP experience in terms of challenges with accessing desired care and coverage

  * Where are families experiencing challenges with accessing desired care and coverage? (drugs, assistive devices, services) Is it different for the different phenotypes of the disease?
  * What is the challenge? (financial, time, stress, others)
  * What is the life impact of that challenge? (work and educational impact, lack or delay of treatment, others)

ELIGIBILITY:
Inclusion Criteria:

* Participant must be a person with Niemann-Pick disease who is 18 years or older or The parent/legal guardian of a person with Niemann-Pick disease. Please note: Parents whose child has passed on are able to participate in the RSVP. Parents whose child has passed on in the last two years are also able to participate in the interview. Please note that only one family member will be eligible to complete the RSVP and interview for one family.
* Confirmed diagnosis of Niemann-Pick disease, confirmed by membership in the NNPDF or by provision of a proof of disease form
* Able to read, write and communicate in English
* Able to grant informed consent
* Willing to complete a survey and RSVP, and to participate in a 30-minute telephone interview
* Ability to view or receive a document from the interviewer before or during the interview (web browser, ability to receive a text, fax or document by mail)

Exclusion Criteria:

- Inability to meet any of the above 6 criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Within the United States, patients or the parent/caregiver of patients who have been diagnosed with any of the 7 known subtypes of Niemann-Pick disease
Sampling Method: Non-Probability Sample
Enrollment: 76 (Actual)
Dates: Start 2020-06-15 (Actual); Primary Completion 2020-09-21 (Actual); Study Completion 2020-09-21 (Actual)

PRIMARY OUTCOMES:
Health Insurance Literacy | July 2020- September
  Health insurance literacy will be measured by a score on a brief quiz regarding health insurance key terms as well as self-ratings regarding various aspects of the participants' ability to navigate and understand insurance
Health Insurance Coverage | July 2020- September
  Health insurance coverage will be measured by the different multiple choice and open-ended questions based on the services available under the participants' insurance plan as well as their reported difficulty with navigating their plan and obtaining what they need for Niemann-Pick

CONTACTS AND LOCATIONS:
Overall Officials: George A Diaz, MD, PhD, Principal Investigator — Icahn School of Medicine at Mount Sinai; Justin Hopkin, MD, Study Chair — National Niemann-Pick Disease Board Chair
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The data for each question in the study will be analyzed and reported by Engage Health using descriptive statistics as appropriate for the nature of the data collected-frequency distributions, cross tabulations and measures of central tendency and dispersion.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: September 2020